CLINICAL TRIAL: NCT02621593
Title: Feasibility of Intense Pulsed Light (IPL) for Reducing Dry Eye Symptoms Caused by Meibomian Gland Dysfunction (MGD)
Brief Title: Feasibility of IPL for Reducing Dry Eye Symptoms Caused by MGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-VBU-M22-15-01
Record Dates: First submitted 2015-11-24; First posted 2015-12-03 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Dry Eye Syndromes
Keywords: Meibomian Gland Dysfunction; Dry eye symptoms; Intense Pulsed Light
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment of dry eye secondary to MGD (Experimental): Intervention: Treatment of dry eye symptoms secondary to MGD with the M22-IPL system
  Interventions: Device: M22-IPL

INTERVENTIONS:
Device: M22-IPL — The IPL hand piece operates at a spectrum of 400-1200nm with 7 different filters that can be easily inserted to the hand piece to treat different conditions. The IPL hand piece also includes 2 different sapphire cooled light guides of 8x15mm and 15x35mm. The cut-off filters that will be used for this evaluation are filters blocking wavelengths of 560 and 595 nm.

SUMMARY:
The purpose of this study is to evaluate if, in patients with meibomian gland dysfunction (MGD), treatment with the Lumenis M22 Intense Pulsed Light (IPL) system causes a reduction in dry eye symptoms post-treatment, compared to pre-treatment.

DETAILED DESCRIPTION:
The IPL module has FDA clearance (K142860) for a wide range of indications, including benign cavernous hemangiomas, benign venous malformations, telangiectasia, port-wine stains, pigmented lesions and erythema of rosacea. As shown by a retrospective study, in over 85% of the cases, using IPL in subjects with ocular rosacea also alleviated the symptoms of DED caused by MGD. No serious adverse events were recorded, suggesting that IPL therapy administered close to the ocular orbits is safe (provided that the eyes are shielded). However, the above mentioned study was retrospective. Therefore, additional evidence is needed in order to substantiate the hypothesis that alleviation of MGD symptom was facilitated by IPL treatments.

The aim of the current study is to assess the safety and efficacy of IPL treatment for reducing the symptoms of dry eye disease (DED) in subjects with MGD. The study hypothesis is that in a study population of subjects diagnosed with moderate to severe MGD, 4 sessions of IPL therapy with the M22 system, followed by expression of the MGs, will cause a significant increase in tear break-up time post-treatment, compared to pre-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and sign an Informed Consent (IC) form
2. 18-80 years of age
3. Fitzpatrick skin type 1-4
4. Able and willing to comply with the treatment/follow-up schedule and requirements
5. At least 5 non-atrophied glands on each eye's lower eyelid
6. Current diagnosis of moderate to severe MGD in both eyes, including 2 of the following 5 criteria:

   * Tear break-up time (TBUT) ≤ 10 seconds in both eyes;
   * Meibomian gland (MG) score (using the Abbreviated MGD grading system for clinical trials) ≥ 11 in both eyes
   * Corneal Fluorescein Staining (CFS) score (using the Baylor grading scheme) ≥ 10 in both eyes;
   * Tear Osmolarity ≥ 310 milliosmol/L in both eyes, or a difference higher than 8 milliosmol/L between the two eyes
   * SPEED ≥ 10
7. Women of child-bearing age are required to be using a reliable method of birth control (such as an intrauterine device, birth control pills, condom with spermicidal, Nuvaring and partner with vasectomy or abstinence) at least 3 months prior to enrollment and throughout the course of the study.

Exclusion Criteria:

1. Contact lens wearer within the past 1 month and throughout the study
2. Recent ocular surgery or eyelid surgery within the past 6 months
3. Neuro-paralysis in the planned treatment area within the past 6 months
4. Other uncontrolled eye disorders affecting the ocular surface
5. Current use of punctal plugs
6. Pre-cancerous lesions, skin cancer or pigmented lesions in the planned treatment area
7. Uncontrolled infections or uncontrolled immunosuppressive diseases
8. Subjects who have undergone laser in situ keratomileusis (LASIK) surgery within the past 6 months
9. Diseases in the planned treatment area that could be stimulated by light at 560 nm to 1200 nm (e.g., Herpes simplex 1 and 2, Systemic Lupus erythematosus, porphyria)
10. Use of photosensitive medication and/or herbs that may cause sensitivity to 560-1200 nm light exposure, such as Isotretinoin, Tetracycline, or St. John's Wort
11. Over exposure to sun within the past 4 weeks, in the judgment of the treating physician
12. Pregnancy and nursing
13. Administration of prescription eye drops for dry eye within the past 48 hours, excluding artificial tears
14. Radiation therapy to the head or neck within the past year, or planned radiation therapy within 8 weeks after completion of all IPL treatments
15. Treatment with chemotherapeutic agent within the past 8 weeks, or planned chemotherapy within 8 weeks after completion of all IPL treatments
16. New topical treatments within the area to be treated, or oral therapies within the past 3 months, except over-the-counter acetaminophen-based analgesics (such as Extra Strength Tylenol®) for pain management after study treatment
17. Change in dosage of any systemic medication within the past 3 months
18. Anticipated relocation or extensive travel outside of the local study area preventing compliance with follow-up within the next 16 weeks
19. Any condition revealed during the eligibility screening process whereby the physician deems the subject inappropriate for this study
20. Declared legally blind in one eye
21. History of migraines, seizures or epilepsy
22. IPL treatment within the past 12 months
23. Lipiflow treatment, or any equivalent treatment, within the past 12 months
24. Expression of the meibomian glands within the past 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Tear Break-up time in seconds, using the standard Fluorescein staining method | from Baseline to 3 weeks after the 3rd treatment and 3 weeks after the fourth/final treatment
  The number of seconds that elapse between the last blink of the eye to the appearance of the first dry spot in the tear film

SECONDARY OUTCOMES:
Corneal fluorescein staining score, using the Baylor Scheme | from Baseline to 3 weeks after the 3rd treatment; 3 weeks after the fourth/final treatment; 6 weeks after the final treatment
  The cornea will be viewed and logically divided to 5 zones: central, superior, inferior, temporal and nasal. In each of the 5 zones, grading will be as follows: 0 dots = 0; 1-5 dots = 1; 16-30 dots = 3; > 30 dots = 4; One point will be added to the score in case of 1 area of confluent staining. Two points will be added to the score in case of two or more areas of confluent staining. The total score is the sum of scores in the 5 zones
Meibomian gland score, using the "Abbreviated MGD grading system for clinical trials" | from Baseline to 3 weeks after the 3rd treatment; 3 weeks after the fourth/final treatment; 6 weeks after the final treatment
  1. Thickening of the upper lid margin (0-3, where 0 is normal and 3 is severe). A value of at least 1 (mild) is consistent with DED.
  2. Vascularity of the upper lid margin (0-3, where 0 is normal and 3 is severe engorgement). A value of at least 1 (mild engorgement) is consistent with DED.
  3. Number of telangiectasias (0-3, where 0 = none, 1 = single, 2 = two to four and 3 = above four). A value of at least 2 (2-4 telangiectasias) is consistent with DED.
  4. Of the central 10 glands of the upper eyelid- number of plugged glands: a value of at least 2 is consistent with DED. The total score is computed by summing the scores of the 8 categories above.
Subjective symptoms, using the SPEED questionnaire | from Baseline to 3 weeks after the 3rd treatment; 3 weeks after the fourth/final treatment; 6 weeks after the final treatment
  SPEED is a validated questionnaire for quantifying the subjective symptoms of DED. The questionnaire will be filled by the study investigator (with questions answered by the subject). In 4 symptoms are evaluated: (1) dryness, grittiness or scratchiness; (2) Soreness or Irritation; (3) Burning or watering; and (4) Eye fatigue. Two types of questions are asked about these symptoms: frequency and severity.
  In the Frequency questions, subjects evaluate the 4 symptoms above on a 0-3 scale: 0 = Never; 1 = Sometimes; 2 = Often; and 3 = All the time.
  In the Severity questions, subjects evaluate the 4 symptoms above on a 0-4 scale: 0 = No problems; 1 = Tolerable (not perfect but not uncomfortable); 2 = Uncomfortable (irritating but does not interfere with my day); 3 = Bothersome (irritating and interferes with my day); and (4) Intolerable (unable to perform my daily tasks). The total score is the sum of the Frequency answers and the Severity answers.
Tear Osmolarity in milliosmol/liter, using a lab-on-a-chip system to simultaneously collect and analyze the electrical impedance of a tear sample | from Baseline to 3 weeks after the 3rd treatment; 3 weeks after the fourth/final treatment; 6 weeks after the final treatment
  In this current study, tear osmolarity will be measured using a lab-on-a-chip system to simultaneously collect and analyze the electrical impedance of a tear sample (TearLab, San Diego, CA, USA). A small tear sample of 50 nL will be collected from the lower meniscus, using a disposable test chip by passive capillary action, and transferred to the device. Several seconds after the transfer, readings will be given in milliOsmol/L
Lipid Layer Thickness in nanometers, using an interferometer | from Baseline to 3 weeks after the 3rd treatment; 3 weeks after the fourth/final treatment; 6 weeks after the final treatment
  lipid layer thickness will be measured using an interferometer. In interferometry, when white light is projected over the cornea, a color interference pattern is produced due to specular reflection at the lipid-aqueous interface. The reflected colors from the tear film are captured on a high-resolution video. Each recorded pixel is analyzed, and compared with a color progression table. The output is expressed as interference color units (ICUS), which correlate with lipid layer thickness

OTHER OUTCOMES:
Incidence of treatment-related adverse events and serious adverse events | 1 day after baseline; 1 week after baseline ; 3 weeks after baseline (Tx2); 6 weeks after baseline (Tx3); 9 weeks after baseline (Tx4/FU1); 12 weeks after baseline (FU2); and 15 weeks after baseline (FU3)
  Evaluation will be done by subject's report and/or by the physician's judgment
immediate/short term skin response | At Baseline (Tx1); 3 weeks after baseline (Tx2); 6 weeks after baseline (Tx3); and 9 weeks after baseline (Tx4/FU1)
  Evaluation will be done by the physician judgment
Subjective level of pain/discomfort. | At Baseline (Tx1); 3 weeks after baseline (Tx2); 6 weeks after baseline (Tx3); and 9 weeks after baseline (Tx4/FU1)
  Evaluation will be done by the subject, using a Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Dell, MD, Principal Investigator — Medical Director, Dell LAser Consultants
Locations (2):
- United States (2):
  - Gaster Eye Center, Beverly Hills, California
  - Dell Laser Consultants, Austin, Texas